CLINICAL TRIAL: NCT04350307
Title: Differential Rates of Intravascular Uptake and Pain Perception During Lumbosacral Transforaminal Epidural Steroid Injection Using a 22-gauge Needle Versus 25-gauge Needle
Brief Title: Comparison of Intravascular Uptake and Pain Perception During Epidural Injection Using 22 Gauge vs 25 Gauge Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Rothman Institute Orthopaedics (Other)
Responsible Party: Principal Investigator, Robin Raju, DO, Clinical Assistant Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000023982
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Pain; Needle Injury
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This was a prospective single blind randomized clinical trial.
Who Masked: Participant
Masking Description: Randomization was done separately for each provider based on a computer generated algorithm. Patients were blinded to the gauge of the needle used for the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 22-Gauge Arm (Active Comparator): Patient undergoing epidural injection in this arm will get 22-gauge Quincke needle
  Interventions: Device: 22-gauge needle; Device: 25-gauge needle
- 25-Gauge Arm (Active Comparator): Patient undergoing epidural injection in this arm will get 25-gauge Quincke needle
  Interventions: Device: 22-gauge needle; Device: 25-gauge needle

INTERVENTIONS:
Device: 22-gauge needle — 22-gauge Quincke needle used for epidural injection
Device: 25-gauge needle — 25-gauge Quincke needle used for epidural injection

SUMMARY:
The aim of the study was to quantify the difference between a 22-gauge needle and 25-gauge needle during lumbosacral epidural steroid injection in regards to intravascular uptake and pain perception. There is the notion that a smaller gauge needle may lead to less intravascular uptake and less pain.

DETAILED DESCRIPTION:
Inadvertent intravascular injection has been suggested as the most probable mechanism behind serious neurological complications during transforaminal epidural steroid injections. There is the notion that a smaller gauge needle may lead to less intravascular uptake and less pain. The aim of the study was to quantify the difference between a 22-gauge needle and 25-gauge needle during lumbosacral transforaminal epidural steroid injection in regards to intravascular uptake and pain perception.

ELIGIBILITY:
Inclusion Criteria:

1. patients with low back pain and/or radicular pain,
2. patients scheduled for lumbosacral TFESI.

Exclusion Criteria:

1. patients with contrast/local anesthetic allergy,
2. patients with pregnancy, coagulopathy, systemic infection, and inability to provide informed consent,
3. vulnerable patient population including prisoners,
4. patients with severe anxiety,
5. patients with prior lumbar surgery,
6. age <18 years old, and
7. Body Mass Index (BMI) > 40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Raju, DO, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raju R, Mehnert M, Stolzenberg D, Simon J, Conliffe T, Gehret J. Differential rates of intravascular uptake and pain perception during lumbosacral epidural injection among adults using a 22-gauge needle versus 25-gauge needle: a randomized clinical trial. BMC Anesthesiol. 2020 Sep 3;20(1):222. doi: 10.1186/s12871-020-01137-0. PMID 32883241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 22-Gauge Arm | 25-Gauge Arm
Started | 84 | 78
Completed | 84 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 22-Gauge Arm | 25-Gauge Arm | Total
Number analyzed (Participants) | 84 | 78 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 20 | 44
  >=65 years | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (2) | 57 (3) | 58 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 37 | 83
  Male | 38 | 41 | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 84 | 78 | 162

OUTCOME MEASURES:

1. Primary Outcome: Intravascular Uptake
Description: The intravascular uptake percentage reported in the study is the percent of 'needles' that showed intravascular uptake. Hence higher 'intravascular uptake percentage' means worse outcome. The mean percentages were averaged across participants were compared between treatment arms.
  Presence or absence of intravascular uptake during live fluoroscopy and/or blood aspiration per needle. Once needle reached its target (epidural space), contrast was injected to confirm the presence or absence of intravascular uptake via live fluoroscopy or aspiration was attempted using a syringe to confirm the presence or absence of intravascular uptake. If contrast pattern suggested needle was in a vessel or blood was aspirated using a syringe, outcome measure was marked 'PRESENT'. If contrast pattern suggested needle was not in a vessel and no blood was aspirated using a syringe, outcome measure was marked 'ABSENT'. In other words, primary outcome measure was binary in nature.
Time Frame: During the procedure
Measure: Mean (95% Confidence Interval); unit: percentage of total number of needle
Arm/Group | 22-Gauge Arm | 25-Gauge Arm
Number analyzed (Participants) | 84 | 78
percentage of total number of needle | 5.9 [1.9 to 9.8] | 7.1 [2.4 to 11.8]

2. Secondary Outcome: Patient Reported Pain
Description: Patient reported pain during the procedure (on initial needle entry) on the numerical rating scale (NRS 1-10). Higher numbers implies higher severity of pain. Lower numbers implies lower severity of pain
Time Frame: During the procedure
Population: Average NRS during the initial needle entry
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 22-Gauge Arm | 25-Gauge Arm
Number analyzed (Participants) | 84 | 78
score on a scale | 3.46 [2.94 to 3.98] | 3.13 [2.57 to 3.69]

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events within 1 month after the injection date.
Arm/Group | 22-Gauge Arm | 25-Gauge Arm
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/78
Other Adverse Events (participants affected / at risk) | 0/84 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04350307/Prot_SAP_002.pdf
  • Informed Consent Form (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT04350307/ICF_003.pdf